CLINICAL TRIAL: NCT05631795
Title: ALPelisib INdia Safety STudy (ALPINIST): A Phase IV, Prospective, Multicenter, Open-label, Non-comparative, Interventional Study to Assess the Safety of Alpelisib Plus Fulvestrant, in Men and Post-menopausal Women With HR Positive, HER2-negative, Advanced Breast Cancer (aBC) With a PIK3CA Mutation, Whose Disease Has Progressed on or After Endocrine Based Treatment.
Brief Title: Study to Assess the Safety of Alpelisib Plus Fulvestrant, in Men and Post-menopausal Women With HR-positive, HER2-negative, Advanced Breast Cancer (aBC) With PIK3CA Mutation, Whose Disease Progressed on or After Endocrine Treatment
Acronym: ALPINIST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBYL719CIN01
Record Dates: First submitted 2022-11-21; First posted 2022-11-30 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Advanced Breast Cancer
Keywords: HR+; HER2-negative; PI3K; CDK4/6 inhibitor; ER+; PgR+; men; postmenopausal; aromatase inhibitor
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1 | interventions — Alpelisib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alpelisib + fulvestrant (Experimental): Alpelisib 300 mg orally once daily starting on Cycle 1 Day 1 in combination with fulvestrant (intramuscular injection) 500 mg on Cycle 1 Day 1 and Day 15, and Day 1 of every cycle thereafter in a 28 day cycle.
  Interventions: Drug: Alpelisib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Alpelisib — Film coated tablet for oral use. Participants will be treated with 300 mg of alpelisib once daily starting on Cycle 1 Day 1
Drug: Fulvestrant — Injection for intramuscular administration. Participants will be treated with fulvestrant 500 mg on Cycle 1 Day 1 and Day 15, and Day 1 of every cycle thereafter in a 28-day cycle.

SUMMARY:
The purpose of this study is to determine the safety of alpelisib plus fulvestrant in men and post-menopausal women with HR-positive, HER2-negative, advanced or metastatic breast cancer (aBC) with a PIK3CA mutation, whose disease has progressed on or after endocrine-based treatment

DETAILED DESCRIPTION:
This is a Phase IV, prospective, multicenter, open-label, non-comparative interventional study to assess the safety of alpelisib plus fulvestrant in men and post-menopausal women with HR-positive, HER2-negative, aBC with a PIK3CA mutation, whose disease has progressed on or after endocrine-based treatment.

Participants will be treated with alpelisib 300 mg orally once daily starting on Cycle 1 Day 1 in combination with fulvestrant (intramuscular injection) 500 mg on Cycle 1 Day 1 and Day 15, and Day 1 of every cycle thereafter in a 28 day cycle. Patients may be discontinued from treatment earlier due to unacceptable toxicity, disease progression, withdrawal of consent, or at the discretion of the investigator or the patient.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with confirmed PIK3CA mutant advanced or metastatic breast cancer
* Postmenopausal females and males ≥ 18 years old with confirmed HR-positive, HER2-negative advanced or metastatic breast cancer.
* Adequate liver function
* Adequate renal function
* Fasting plasma glucose (FPG) ≤140 mg/dL (7.7 mmol/L) and glycosylated hemoglobin (HbA1c) ≤ 6.4%
* ECOG (Eastern Cooperative Oncology Group) Performance Status < 2
* Fasting Serum amylase ≤ 2 × ULN and Fasting Serum lipase ≤ ULN
* Potassium within normal limits, or corrected with supplements
* Calcium (corrected for serum albumin) and magnesium within normal limits or ≤ grade 1 if judged clinically not significant by the investigator

Key Exclusion Criteria:

* Known hypersensitivity to alpelisib or fulvestrant, or to any of the excipients of alpelisib or fulvestrant
* Participant ineligible for endocrine therapy per the investigator's judgment
* Participant has received prior treatment with any PI3K inhibitors and / or mTOR inhibitor
* Participant with type I diabetes or not controlled type II (based on FPG and HbA1c, see inclusion criterion 6)
* Participant has a concurrent malignancy or malignancy within 3 years of study screening period, with the exception of adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer
* Participant has not recovered to grade 1 or better from related side effects of prior anti cancer therapy (with the exception of alopecia)
* Participants receiving concomitant immunosuppressive agents or chronic corticosteroids use at the time of study entry except in cases outlined below: Topical applications, inhaled sprays, eye drops or local injections are allowed. Participants on stable low dose of corticosteroids for at least two weeks prior to enrollment are allowed
* Bilateral diffuse lymphangitic carcinomatosis
* Participants with a known history of HIV seropositivity. Screening for HIV infection at baseline is not required
* Active, bleeding diathesis, or on oral anti-vitamin K medication (except low dose warfarin and acetylsalicylic acid or equivalent, as long as the INR is ≤2.0)
* Any severe and/ or uncontrolled medical conditions
* Participant with severe liver impairment (Child Pugh score B/C)
* Participant has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs
* Participant has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, contraindicate patient participation in the clinical study
* Participant has documented pneumonitis/interstitial lung disease which is active and requiring treatment
* Participant has active cardiac disease or a history of cardiac dysfunction
* Participants with unresolved osteonecrosis of the jaw
* Participant has a history of severe cutaneous reactions like Stevens-Johnson-Syndrome (SJS), Erythema Multiforme (EM), Toxic Epidermal Necrolysis (TEN), or Drug Reaction with Eosinophilia and Systemic Symptoms (DRESS).
* Participant is a nursing (lactating) or pregnant woman
* Participant is a woman of child-bearing potential defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during study treatment and at least for 1 week (for alpelisib) or 1 year (for fulvestrant based on prescribing label) after the last dose of each study drug (whichever comes later).
* Participant is a sexually active male unwilling to use a condom during intercourse while taking study treatment, and for 1 week (for alpelisib) or 1 year (for fulvestrant based on prescribing label) after stopping each study drug (whichever comes later). A condom is required for all sexually active male participants to prevent them from fathering a child AND to prevent delivery of study treatment via seminal fluid to their partner. In addition, male participants must not donate sperm during study and up to the time period specified above.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with at least one on-treatment adverse events (AEs) | From start of treatment up to 30 days after last dose of study treatment, assessed up to approximately 7 months
  Percentage of participants with at least one on-treatment AEs. An AE is any untoward medical occurrence (an unfavourable/unintended sign - including an abnormal laboratory finding), symptom, or disease) in a participant.
  On-treatment period is defined as up to 30 days after last dose of study drug

SECONDARY OUTCOMES:
Percentage of participants with Serious AEs (SAEs) | From start of treatment up to 30 days after last dose of study treatment, assessed up to approximately 7 months
  Percentage of participants with SAEs. An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, or is an abnormal pregnancy outcome
Percentage of participants with Adverse Drug Reactions (ADRs) | From start of treatment up to 30 days after last dose of study treatment, assessed up to approximately 7 months
  Percentage of participants with ADRs. An ADR is defined as AEs that are, in the investigator's opinion, of causal relationship to the study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- India (12):
  - Novartis Investigative Site, Guwahati, Assam
  - Novartis Investigative Site, Surat, Gujarat
  - Novartis Investigative Site, Thalassery, Kerala
  - Novartis Investigative Site, Trivandrum, Kerala
  - Novartis Investigative Site, Bhopal, Madhya Pradesh
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Ahmedabad
  - Novartis Investigative Site, Kolkata

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com